CLINICAL TRIAL: NCT05941312
Title: Clinical and Radiographic Evaluation of the Use of Different Autologous Products in the Treatment of Periodontal Intrabony Defects
Brief Title: Different Autologous Products in The Treatment of Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ahmet Cemil Talmac, PhD,DDA, Assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17.06.2020/19
Record Dates: First submitted 2023-06-14; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Periodontal Pocket
Keywords: Autologous bone graft; concentrated growth factor; platelet-rich fibrin
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CONTROL GROUP (GROUP 1) (Active Comparator): Only open flap debridement (OFD):
  Conventional OFD surgery was applied to patients in all groups which began with local anesthesia (4% articaine with 1:100 000 epinephrine) after the surgical area was disinfected. Defects were thoroughly debrided firstly by using periodontal curettes and then cleaned by piezoelectric ultrasonic scaler. For the control group, the defects were left without adding any products.
  Interventions: Procedure: autologous products
- GROUP 2 (Active Comparator): Conventional OFD surgery was applied to patients in all groups which began with local anesthesia (4% articaine with 1:100 000 epinephrine) after the surgical area was disinfected. Defects were thoroughly debrided firstly by using periodontal curettes and then cleaned by piezoelectric ultrasonic scaler. After the operation area was washed thoroughly with saline, platelet-rich fibrine (PRF) was placed inside defects
  Interventions: Procedure: autologous products
- GROUP 3 (Active Comparator): Conventional OFD surgery was applied to patients in all groups which began with local anesthesia (4% articaine with 1:100 000 epinephrine) after the surgical area was disinfected. Defects were thoroughly debrided firstly by using periodontal curettes and then cleaned by piezoelectric ultrasonic scaler. After the operation area was washed thoroughly with saline, Consantrated Growth Factor (CGF) was placed inside defects
  Interventions: Procedure: autologous products
- GROUP 4 (Active Comparator): Conventional OFD surgery was applied to patients in all groups which began with local anesthesia (4% articaine with 1:100 000 epinephrine) after the surgical area was disinfected. Defects were thoroughly debrided firstly by using periodontal curettes and then cleaned by piezoelectric ultrasonic scaler. After the operation area was washed thoroughly with saline, autologous bone graft (ABG) was placed inside defects
  Interventions: Procedure: autologous products

INTERVENTIONS:
Procedure: autologous products — After the operation area was washed thoroughly with saline, autologous products were placed inside defects according to the related group. For the control group, the defects were left without adding any products.

SUMMARY:
The aim of this study is to evaluate and compare the efficiencies of platelet-rich fibrin (PRF), concentrated growth factor (CGF) and autologous bone graft (ABG) in the treatment of patients who have intrabony pockets clinically and to assess the alveolar bone gain (AB gain) radiographically ((Panoramic X-ray and cone-beam computed tomography (CBCT) X-ray)).

DETAILED DESCRIPTION:
Periodontitis is a complex multifactorial inflammatory disorder of periodontium, which occurs due to accumulations of microorganism that lead to gradual damage of periodontal tissues resulting in the creation of periodontal defects and recession of gingiva. This leads to the initiation of bone resorption forming bone defect known as periodontal pocket (PP). PP could be treated by surgical and non-surgical procedures. Non-surgical treatment or initial periodontal treatment (IPT) aims to remove irritant factors of periodontal disease. Surgical procedure has to be applied if inflammation persists after non-surgical procedures. One of the most common surgical procedures used for treatment of PP is an open flap debridement (OFD) which aims to remove infection and inflamed tissue, and to establish the appropriate biological situations essential for periodontal regeneration. However, the regeneration of tissues damaged by periodontitis could not be accomplished by OFD alone. Some autologous products that can be used in regenerative periodontal treatment include: ABG, autologous soft tissue graft and autologous platelet concentrates (APC).

ABGs consist of live osteoblasts, osteoprogenitor stem cells and all the three components for tissue engineering, i.e, scaffold, cells, and signaling molecules. Among the several available regeneration substances, only ABG involves osteoconductive, osteoinductive, and osteogenic properties. Due to their favorable characteristics, ABGs have been regarded as the "gold standard", and the most successful material that can be used in periodontal regeneration surgery. Despite being quite effective, ABGs have some drawbacks, including limited donor locations, insufficient bone amount, another site surgery, the possibility of some unexpected bone resorption and donor site morbidity, which includes pain, infection, sensory loss, and bleeding. Because of these shortcomings, the use of other autologous products such as autologous platelet concentrates (APC ; PRF, CGF) has become needed.

PRF is a second-generation autologous platelet concentrate as it is a natural concentrate prepared directly by taking blood from the patient without adding any anticoagulant. PRFs were firstly introduced in 2001 with the aim of simplifying the platelet-rich plasma (PRP) preparation protocol and overcoming its drawbacks. It is inexpensive, time saving, and it does not require chemical alteration in collected blood. Literature showed that the PRF membrane could stay intact and release continuously large quantities of growth factors slowly for at least 1 week, due to its fiber network scaffold. PRF shows effective outcomes in the surgical management of periodontal intra-bony and furcation defects which lead to noticeable improvement of PD and CAL. Some other dental applications are socket preservation after extraction, root covering procedure, third-molar surgery, alveolar ridge preservation, guided tissue regeneration and sinus elevation. Furthermore, PRF has the ability to enhance osseointegration of implants and can be used with grafting materials as natural resorbable membrane as an alternative to collagen membrane in managing periodontal and peri-implant defects. Nevertheless, the PRF membrane has fast biodegradability (up to 14 days). However, PRF has some limitation, as it required to be used as quickly as possible after preparation. Recently, researchers developed new products of the PRF that aim to improve the properties of PRF and obtain a better autogenous biological material by changing the centrifuge time and speed (Injectable-PRF, Advanced-PRF and CGF).

CGF is an advanced second-generation platelet concentrate, which consists of diverse growth factors that stimulate and accelerate bone formation and soft and hard tissue healing. CGF can also improve the quality of the produced new bone. CGF was firstly introduced by Sacco in 2006 as a recent improved formulation of PRF which contains high amount of growth factors and can be used successfully in regenerative treatments. It has a different preparation protocol by alternating and controlling centrifugation speeds manually or by using a special centrifuge machine, which permits the formation of a considerably larger and firmer fibrin matrix which is more abundant in growth factors compared to those observed in PRP and classic PRF. He et al26 reported that the three-dimensional fiber network scaffold of CGF could help in releasing growth factors gradually for a period between 7-10 days.

So, according to recent findings in the literature, the hypothesis of this study was that the treatment of periodontal intrabony defects by using OFD in combination with autologous products (PRF, CGF and ABG) would lead to effective outcomes compared to OFD alone. Therefore the aim of this randomized controlled clinical study was to evaluate the effects of different autologous products (PRF, CGF and ABG) on the treatment of periodontitis patients who have intrabony pockets and to compare between their efficiency clinically and radiographically.

ELIGIBILITY:
Inclusion Criteria:

1. no systemic disease
2. presence of two-wall intrabony defects with radiographic depth ≥3 mm
3. presence of at least four intrabony defects, one in each quadrant (in molar and premolar regions)
4. pocket depth ≥5mm
5. no periodontal treatment within past 6 months

Exclusion Criteria:

1. Smoking
2. Having a systemic disease that may affect the treatment results such as uncontrolled diabetes, metabolic bone diseases, hematological disorders, radiotherapy in the head and neck region, kidney disease,
3. Being in pregnancy or breastfeeding period,

Ages: 30 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Probing depth (PD) | Baseline (day 0) PD was evaluated. The change between baseline measurements and day 90 measurements was evaluated. Finally, the change between the baseline measurements and the 180th day measurements was evaluated.
  Probing depth (PD) was measured from the gingival margin to the bottom of the pocket
Alveolar bone height loss (ABHL) | Baseline (day 0) ABHL was evaluated. The change between the baseline measurements and the 180th day measurements was evaluated.
  Alveolar bone height loss (ABHL) was measured using CBCT images from the distance between cementoenamel junction to the most apical base of the pocket.

SECONDARY OUTCOMES:
Plaque index (PI) | days 0, 30, 90 and 180
  PI was measured from the all diseased teeth. The PI score was calculated with Silness-Loe plaque index.
  0:absence of microbial plaque
  1. Thin film of microbial plaque along the free gingival margin
  2. moderate accumulation with plaque in the sulcus
  3. large amount of plaque in sulcus or pocket along the free gingival margin
Gingival index (GI) | days 0, 30, 90 and 180
  GI was measured from the all diseased teeth. The GI score was calculated with Silness-Loe plaque index.
  0:Normal gingiva
  1. Mild inflammation: slight change in color, slight oedema, no bleeding on probing
  2. Moderate inflammation: redness,oedema and glazing, bleeding on probing
  3. Severe inflammation: marked redness and oedema, ulceration, tendency to spontaneous bleeding
Tooth mobility (TM) | days 0, 30, 90 and 180
  The tooth mobility (TM) by using Periotest M device
Clinical attachment level (CAL) | days 0, 90 and 180
  The clinical attachment level (CAL) was measured from the cementoenamel junction (CEJ) to the deepest point in the pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Basem ALSHUJAA, PhD, Principal Investigator — Special dental clinic; Ahmet Cemil TALMAC, PhD, Study Director — Yuzuncu Yil University; Dicle ALTINDAL, PhD, Study Chair — Yuzuncu Yil University; Anas ALSAFADI, PhD, Study Chair — Special dental clinic; Abdullah Seckin ERTUGRUL, PhD, Study Chair — Izmir Katip Celebi University
Locations (1):
- Ahmet Cemil TALMAC, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghanaati S, Booms P, Orlowska A, Kubesch A, Lorenz J, Rutkowski J, Landes C, Sader R, Kirkpatrick C, Choukroun J. Advanced platelet-rich fibrin: a new concept for cell-based tissue engineering by means of inflammatory cells. J Oral Implantol. 2014 Dec;40(6):679-89. doi: 10.1563/aaid-joi-D-14-00138. PMID 24945603